CLINICAL TRIAL: NCT02130518
Title: A Multicenter, Randomized, Double-Blind, Efficacy Study of Auriclosene Irrigation Solution on Indwelling Urinary Catheter Patency
Brief Title: Efficacy Study of Auriclosene Irrigation Solution on Urinary Catheter Patency
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NovaBay Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CL1401
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Urinary Catheter Blockage and Encrustation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auriclosene (AIS) (Experimental): Auriclosene Irrigation Solution, 0.2%, 8 treatments over 4 weeks
  Interventions: Drug: Auriclosene Irrigation Solution, 0.2%
- Auriclosene Vehicle Solution (Placebo Comparator): Auriclosene Vehicle Solution, 8 treatments over 4 weeks
  Interventions: Drug: Auriclosene Vehicle Solution

INTERVENTIONS:
Drug: Auriclosene Irrigation Solution, 0.2%
  Arms: Auriclosene (AIS)
Drug: Auriclosene Vehicle Solution
  Arms: Auriclosene Vehicle Solution

SUMMARY:
Long-term indwelling urinary catheters are associated with chronic recurrent urinary tract infections and blockage caused by crystalline biofilm accumulation (encrustation) of the catheter surfaces. When the urine and catheter are colonized by urease-producing bacteria such as Proteus mirabilis, encrustation of the catheter is likely to occur.

The use of a catheter irrigation solution that can prevent biofilm formation and encrustation leading to blockage may keep the catheter patent longer, resulting in fewer catheter changes, potentially lower incidence of UTIs and better patient quality of life.

Auriclosene is a non-antibiotic, fast-acting, broad-spectrum antimicrobial, which exhibits potential for the rapid decolonization of a range of urologic pathogens, including the urease-producing Proteus mirabilis.

Subjects will be randomized to either Auriclosene Irrigation Solution or Auriclosene Vehicle solution.

ELIGIBILITY:
Inclusion Criteria:

* Subject requiring an indwelling urinary catheter with a history of catheter blockage and/or encrustation
* Screening within 30 days of randomization

Exclusion Criteria:

* Systemic antibiotic use within 14 days of first treatment
* Investigational drug or device within 30 days if enrollment
* Current infection requiring treatment with systemic antibiotics
* Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Percent flow rate reduction of study catheters at time of removal | Up to 29 Days

SECONDARY OUTCOMES:
Number of study catheters removed due to clinical catheter blockage | Up to 29 days
Number of subjects with serious and non-serious adverse events | Up to 29 Days

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Najafi-Tagol, MD, Study Director — NovaBay Pharmaceuticals, Inc.
Locations (17):
- United States (17):
  - Los Amigos Research and Education Institute, Downey, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Chesapeake Urology Research Associates, Owings Mills, Maryland
  - Lahey Hospital and Medical Clinic, Burlington, Massachusetts
  - Urology Center Research Institute, Englewood, New Jersey
  - Delaware Valley Urology, LLC, Voorhees Township, New Jersey
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - Urology Group of New Mexico, Albuquerque, New Mexico
  - The Urological Institute of Northeastern NY, Albany, New York
  - McKay Urology, Charlotte, North Carolina
  - Eastern Urological Associates, Greenville, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Great Lakes Medical Research, Mentor, Ohio
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Dean Clinic, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin